CLINICAL TRIAL: NCT05541016
Title: DART 2.0: ctHPV-DNA Informed De-Escalated Adjuvant and Definitive Radiation Therapy
Brief Title: De-Escalated Adjuvant and Definitive Radiation Therapy Informed by DART 2.0 ctHPV-DNA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMROR2271; NCI-2022-06932 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-004443 (Other: Mayo Clinic in Rochester); DART 2.0 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2022-08-30; First posted 2022-09-15 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Clinical Stage I HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Human Papillomavirus-Related Oropharyngeal Squamous Cell Carcinoma; Stage I Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage II Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms; Carcinoma | interventions — Specimen Handling; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Docetaxel; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy; Observation; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Group 1 (observation) (Active Comparator): Patients undergo observation following standard of care surgery. Patients undergo modified barium swallow study (MBSS) at pre-op, 2 weeks post-op, and 3 months follow-up. Patients also undergo CT, PET/CT, or magnetic MRI at baseline and 3 months and 1, 2 and 5 years post treatment. Patients undergo blood specimen collection for NavDx testing at pre-op, 1-2 days post-op, 2 weeks post-op, and 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 48, and 60 months as well as saliva sample collection at pre-op, end of RT, and any clinical recurrence.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Modified Barium Swallow Study; Other: Observation Activity; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire
- Group 2 (DART, docetaxel) (Experimental): Patients undergo DART with/without mucosal sparing BID on days 1-12 Monday-Friday for a total of 20 fractions within 8 weeks of standard of care surgery. Patients receive concurrent docetaxel IV over 1 hour on days 1 and 8 (Mondays preferred). Treatment continues in the absence of disease progression or unacceptable toxicity. Patients undergo MBSS at pre-op, 2 weeks post-op, and 3 and 12 months post-treatment. Patients also undergo CT, PET/CT, or MRI at baseline and 3 months and 1, 2 and 5 years post treatment. Patients undergo blood specimen collection for NavDx testing at pre-op, 1-2 days post-op, 2 weeks post-op, end of RT, and 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 48, and 60 months as well as saliva sample collection at pre-op, end of RT, and any clinical recurrence.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Radiation: Diffusing Alpha-emitter Radiation Therapy; Drug: Docetaxel; Procedure: Magnetic Resonance Imaging; Procedure: Modified Barium Swallow Study; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire
- Group 3 (IMRT/IMPT, with/without cisplatin) (Experimental): Patients undergo IMRT or IMPT QD on days 1-40 Monday-Friday for a total of 30 fractions within 6 weeks of standard of care surgery. Depending on risk status, patients may also receive concurrent cisplatin IV over 1-2 hours once a week QW on Monday, Tuesday, or Wednesday or once every 3 weeks for 6 doses (or accepted alternate regimen when drug shortage applies per physician discretion). Treatment continues in the absence of disease progression or unacceptable toxicity. Patients undergo MBSS at pre-op, 2 weeks post-op, and 3 and 12 months post-treatment. Patients also undergo CT, PET/CT, or MRI at baseline and 3 months and 1, 2 and 5 years post treatment. Patients undergo blood specimen collection for NavDx testing at pre-op, 1-2 days post-op, 2 weeks post-op, end of RT, and 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 48, and 60 months as well as saliva sample collection at pre-op, end of RT, and any clinical recurrence.
  Interventions: Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Procedure: Intensity-Modulated Proton Therapy; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Modified Barium Swallow Study; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire
- Group 4 (IMRT/IMPT, cisplatin) (Experimental): Patients undergo IMRT or IMPT therapy QD on days 1-40 Monday-Friday for 28 or 35 fractions based on biomarker response along with concurrent cisplatin IV over 1-2 hours QW on Monday, Tuesday, or Wednesday or once every 3 weeks for 6 doses (or accepted alternate regimen when drug shortage applies per physician discretion). Treatment continues in the absence of disease progression or unacceptable toxicity. Patients undergo MBSS prior to RT and at 3 and 12 months post RT. Patients undergo CT, PET/CT, or MRI at baseline and 3 months and 1, 2 and 5 years post treatment. Patients undergo blood specimen collection for NavDx testing pre-RT, 4 weeks into RT, anticipated fraction 20, end of RT, 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 48, and 60 months as well as saliva sample collection at pre-op, end of RT, and any clinical recurrence.
  Interventions: Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Procedure: Intensity-Modulated Proton Therapy; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Modified Barium Swallow Study; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and saliva specimen collection for NavDx testing
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Group 3 (IMRT/IMPT, with/without cisplatin); Group 4 (IMRT/IMPT, cisplatin)
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography; Computerized axial tomography (procedure)
Radiation: Diffusing Alpha-emitter Radiation Therapy — Undergo DART
  Other Names: DaRT
  Arms: Group 2 (DART, docetaxel)
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate; RP 56976; RP-56976
  Arms: Group 2 (DART, docetaxel)
Procedure: Intensity-Modulated Proton Therapy — Undergo IMPT
  Other Names: IMPT
  Arms: Group 3 (IMRT/IMPT, with/without cisplatin); Group 4 (IMRT/IMPT, cisplatin)
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy; Intensity modulated radiation therapy (procedure)
  Arms: Group 3 (IMRT/IMPT, with/without cisplatin); Group 4 (IMRT/IMPT, cisplatin)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; Magnetic resonance imaging (procedure)
Procedure: Modified Barium Swallow Study — Undergo MBSS
  Other Names: MBS; Modified Barium Swallow; VFSS; Videofluoroscopic Swallowing Study
Other: Observation Activity — Undergo observation
  Other Names: OBSERVATION
  Arms: Group 1 (observation)
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; PT; Positron emission tomography (procedure)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire — Ancillary studies
  Other Names: Questionnaire Administration
  Arms: Group 1 (observation); Group 2 (DART, docetaxel); Group 3 (IMRT/IMPT, with/without cisplatin)

SUMMARY:
This phase II trial examines the use of blood-based biomarkers is to help inform decision making for treatment and radiation therapy for patients with human papillomavirus (HPV) positive oropharyngeal squamous cell cancers. The standard treatments for head and neck cancers are radiation therapy with chemotherapy or surgery potentially followed by radiation therapy with or without chemotherapy. Radiation therapy uses high energy rays to kill tumor cells and shrink tumors. Giving chemotherapy along with radiation may kill more tumor cells. However, the cancer can recur or can spread to other parts of the body and all treatments can be associated with side effects. The purpose of this study is to evaluate a blood-based biomarker, using the NavDx testing device, for head and neck cancers in order to see if it can help improve selection of the intensity of treatment in order to best balance the side effects of treatment with the goal of decreasing cancer recurrence. This test could aid in early detection of recurrence and salvage therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To prospectively incorporate circulating tumor human papillomavirus deoxyribonucleic acid (ctHPVDNA) in combination with clinical and pathologic factors to appropriately select patients for treatment intensity.

II. To demonstrate patients traditionally offered adjuvant radiation therapy (RT) but at low risk of treatment failure based on clinical pathologic and post op ctHPVDNA risk factors have an acceptable 1-year progression free survival (PFS) warranting further study. (Favorable Intermediate Risk [GROUP 1]) III. To demonstrate based on clinical, pathologic, and ctHPVDNA risk factors a select population receiving diffusing alpha-emitter radiation therapy (DART) (+ multiple segment radiation therapy [MSRT] where applicable) is associated with acceptable 2 year PFS. (Unfavorable Intermediate Risk [GROUP 2]) IV. To quantify the rate of recurrence as defined by the 2 year PFS in an identified high risk population using the incorporation of ctHPVDNA. (High Risk [GROUP 3]) V. To prospectively use week 4 ctHPVDNA to guide treatment intensity of 56 versus (vs) 70 Gy with concurrent cisplatin to demonstrate 56 Gy with sufficient ctHPVDNA clearance results in an acceptable 2 year PFS. (Chemoradiation Cohort [GROUP 4])

SECONDARY OBJECTIVES:

I. To compare PFS by treatment arm including at landmark timepoints II. To assess the disease-free survival (DFS) in patients that are disease-free post-treatment.

III. To compare overall survival (OS) by treatment arm including at landmark timepoints.

IV. To compare patient reported outcomes (PROS) by treatment arm and modality. V. To evaluate treatment toxicity by Common Terminology Criteria for Adverse Events (CTCAE) criteria as rated by providers across treatment arms.

VI. To define patterns of recurrence by treatment arm. VII. To describe salvage therapy by treatment arm, including the rate, type, and success of salvage treatment.

VIII. To compare functional outcomes by treatment arm based on modified barium swallow study (MBSS) and Functional Oral Intake Scale (FOIS) by treatment arm.

IX. To return to work parameters by treatment arm as assessed by the Work Productivity and Activity Impairment Questionnaire (WPAI).

X. To quantify the costs of return visits for surveillance. XI. To assess end of treatment ctHPVDNA detectability and its association with PFS by comparing patients with detectable versus undetectable end of treatment ctHPVDNA within treatment arms.

XII. To compare outcomes by institution. XIII. To evaluate rates of post operative bleeding, tracheostomy, and readmission with 6 weeks of resection.

XIV. To compare methods of surveillance in diagnosis of recurrence including clinical evaluation, ctHPVDNA testing, and imaging.

XV. To investigate the impact of tobacco and smoking history on recurrence, PFS, and OS.

XVI. To perform a matched analysis of patients by clinical and pathologic risk factors to MC1273, MC1675, and MC Mucosal Sparing (NCT02736786).

CORRELATIVE RESEARCH OBJECTIVES:

I. Will investigate post-op Day 1 or 2 ctHPVDNA detectability as a surrogate for detectability for later post-op timepoints including risk of recurrence rates.

II. Will analyze salivary samples pre-treatment, post-op, and at the time of recurrence to determine whether salivary ctHPVDNA may further inform recurrence risk and surveillance in HPV(+) oropharyngeal squamous cell carcinoma (OPSCC).

III. Will characterize post-operative drain fluid and compare rates of detectability to blood and saliva in order with the aim to determine whether the regional drain represents a separate regional compartment for analysis.

IV. Will prospectively quantify pretreatment imaging for number of involved nodes, radiographic extranodal extension (rENE) as it relates to pathologic findings and risk of recurrence.

V. Will analyze within category of low intermediate, high intermediate, and high-risk patients the percentage of tumor infiltrating lymphocytes (TILs) and association with recurrence as well as differences across treatment groups.

VI. Will assess whether HPV is integrated vs episomal for each patient and the relationship of ctHPVDNA detectability and outcomes.

VII. Will investigate molecular markers on formalin-fixed paraffin-embedded (FFPE) from primary surgical specimens.

OUTLINE: Patients are assigned to 1 of 4 groups.

GROUP I: Patients undergo observation following standard of care surgery. Patients undergo MBSS at pre-operative (pre-op), 2 weeks post-operative (post-op), and 3 months follow-up. Patients also undergo computed tomography (CT), positron emission tomography (PET)/CT, or magnetic resonance imaging (MRI) at baseline and 3 months and 1, 2 and 5 years post treatment. Patients undergo blood specimen collection for NavDx testing at pre-op, 1-2 days post-op, 2 weeks post-op, and 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 48, and 60 months as well as saliva sample collection at pre-op, end of RT, and any clinical recurrence.

GROUP II: Patients undergo DART with/without mucosal sparing twice daily (BID) on days 1-12 Monday-Friday for a total of 20 fractions within 8 weeks of standard of care surgery. Patients receive concurrent docetaxel intravenously (IV) over 1 hour on days 1 and 8 (Mondays preferred). Treatment continues in the absence of disease progression or unacceptable toxicity. Patients undergo MBSS at pre-op, 2 weeks post-op, and 3 and 12 months post-treatment. Patients also undergo CT, PET/CT, or MRI at baseline and 3 months and 1, 2 and 5 years post treatment. Patients undergo blood specimen collection for NavDx testing at pre-op, 1-2 days post-op, 2 weeks post-op, end of RT, and 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 48, and 60 months as well as saliva sample collection at pre-op, end of RT, and any clinical recurrence.

GROUP III: Patients undergo intensity-modulated radiation therapy (IMRT) or intensity-modulated proton therapy (IMPT) once daily (QD) on days 1-40 Monday-Friday for a total of 30 fractions within 6 weeks of standard of care surgery. Depending on risk status, patients may also receive concurrent cisplatin IV over 1-2 hours once a week (QW) on Monday, Tuesday, or Wednesday or once every 3 weeks for 6 doses (or accepted alternate regimen when drug shortage applies per physician discretion). Treatment continues in the absence of disease progression or unacceptable toxicity. Patients undergo MBSS at pre-op, post-op, and 3 and 12 months post-treatment. Patients also undergo CT, PET/CT, or MRI at baseline and 3 months and 1, 2 and 5 years post treatment. Patients undergo blood specimen collection for NavDx testing at pre-op, 1-2 days post-op, 2 weeks post-op, end of RT, and 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 48, and 60 months as well as saliva sample collection at pre-op, end of RT, and any clinical recurrence.

GROUP IV: Patients undergo IMRT or IMPT therapy QD on days 1-40 Monday-Friday for 28 or 35 fractions based on biomarker response along with concurrent cisplatin IV over 1-2 hours QW on Monday, Tuesday, or Wednesday or once every 3 weeks for 6 doses (or accepted alternate regimen when drug shortage applies per physician discretion). Treatment continues in the absence of disease progression or unacceptable toxicity. Patients undergo MBSS prior to RT and at 3 and 12 months post RT. Patients undergo CT, PET/CT, or MRI at baseline and 3 months and 1, 2 and 5 years post treatment. Patients undergo blood specimen collection for NavDx testing pre-RT, 4 weeks into RT, anticipated fraction 20, end of RT, 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 48, and 60 months as well as saliva sample collection at prior to RT, at the end of RT, at any clinical recurrence.

After completion of study treatment, patients are followed up at 4-6 weeks post treatment, every 3 months post-treatment for 2 years, every 6 months for year 3, and annually for years 4 and 5.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION (optional): Provide written informed consent
* Age >= 18 years
* Histological confirmation of squamous cell carcinoma originating from or suspected to be originating from the oropharynx
* Plan for gross total surgical resection via trans oral surgery with curative intent and at least unilateral neck dissection OR chemoradiotherapy with cisplatin. Note: The patient must be cisplatin eligible even if an alternate is used due to drug shortage
* Absence of distant metastases on standard diagnostic work-up =< 16 weeks prior to registration. (Chest CT or PET/CT)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 1
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing to provide blood samples for correlative research purposes, including anonymous shipment of samples to for NavDx testing

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV)+
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 5 years prior to registration. EXCEPTIONS: Nonmelanotic skin cancer or carcinoma-in-situ of the cervix, or prostate or localized endometrioid endometrial cancer. NOTE: If there is a history or prior malignancy, they must not be receiving other specific treatment for their cancer
* Prior history of radiation therapy to the affected site
* Prior systemic chemotherapy in the last 5 years
* Contraindication to radiation therapy as determined by the treating team
* History of allergic reaction to docetaxel
* Receiving any medications or substances which in the opinion of the investigators would interfere with treatment. Examples could include strong inhibitors of cytochrome P450 3A4 (CYP3A4) at oncologist discretion
* Severe pre-existing ototoxicity or neuropathy that would, in the opinion of the investigator, preclude the use of cisplatin chemotherapy
* cT4 primary tumor

  * NOTE: Patients with no intermediate risk factors after surgery, low risk patients, as defined by T1, T2, tumors with lymph node less than 3cm, no intermediate or high-risk factors such as lymphatic invasion (LVSI), extranodal extension (ENE), perineural invasion (PNI), positive margin, will be withdrawn from study and be observed per current clinical standard of care. Patients found to be both HPV negative and p16 negative will be withdrawn from study.
  * Patients found to have HPV non 16 type, or HPV detectability in blood less than <20tumor tissue modified viral (TTMV) will not be candidates for de-escalation in Groups 1 and 2 and will be treated in Group 3 unless otherwise meeting criteria for low risk. They will receive 60 Gy +/- cisplatin or acceptable alternate regimen when drug shortages of cisplatin exist. If treated primarily with chemoradiation (chemoRT) (Group 4), these patients will not be candidates for de-escalation if TTMV is < 50 TTMV but can remain on study receiving 70 Gy with all corresponding correlative studies applying
  * Patients with unknown (radiologic/clinically occult) primaries but neck adenopathy suspected to be HPV associated oropharyngeal carcinoma can be registered to go on study for Groups 1-3. Should after primary resection, no primary tumor be identified, the patient will be withdrawn from study and be treated per institutional standard of care. Group 4 patients must have an identifiable (clinically or radiologically apparent) primary tumor
  * All treatment primarily, including surgery and chemotherapy will be performed at the enrolling institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From registration to the first of either disease progression/recurrence or death, assessed up to 5 years
  Progression-free survival (PFS), the time from treatment initiation until disease progression or worsening. PFS at specific timepoints will be estimated using Kaplan-Meier methodology.

SECONDARY OUTCOMES:
Progression-free survival (PFS) follow-up | At years 1, 2, 3, 4, and 5
  Progression-free survival (PFS) is defined as the time from treatment initiation until disease progression or worsening. Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response versus (vs.) no response), we'll use logistic regression models.
Disease-free survival (DFS) | From time of surgery and also from end of all treatment across all the groups, assessed up to 5 years
  Disease-free survival (DFS) is the measure of time after treatment during which no sign of cancer is found. Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Overall survival (OS) | At years 1, 2, 3, 4, and 5
  Overall survival (OS) is defined as the duration of patient survival from the time of treatment initiation. Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Patient reported outcomes (PROs) | Up to 5 years
  Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Incidence of adverse events | Up to 5 years
  Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Patterns of recurrence and rate of salvage therapy for Low Intermediate Risk (GROUP 1) and multiple segment radiation therapy (MSRT) + de-escalated adjuvant radiation therapy (DART) | Up to 5 years
  Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Functional outcomes - modified barium swallow study (MBSS) | Up to 5 years
  Measured by modified barium swallow (MBSS). Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Functional outcomes - PROs | Up to 5 years
  Measure by patient reported outcomes (PROs). Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Proton vs photon treatment toxicity - PROs | Up to 5 years
  Assessed by PROs. Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Proton vs photon treatment toxicity - MBSS | Up to 5 years
  Assessed by MBSS. Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Proton vs photon treatment toxicity - dosimetric differences | Up to 5 years
  Assessed by dosimetric differences including to organs at risk and the primary tumor bed in the case of mucosal sparing. Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Costs of return visits for surveillance | Up to 5 years
  Presented descriptively and ANOVA models with tukey's adjustment for pairwise comparison will be utilized to test difference in arms.
Assessment of surveillance circulating human papillomavirus deoxyribonucleic acid (ctHPVDNA) preceding clinical or radiologic detection of recurrence | Up to 5 years
  Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Matched analysis of patients by clinical and pathologic risk factor to MC1273 and MC1675 de-escalation arms to overall GROUP 1 and GROUP 2 cohorts including 2-year PFS | Up to 5 years
  Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Evaluation of return to work | Up to 5 years
  Will be assessed by the Work Productivity and Activity Impairment Questionnaire (WPAI). Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Evaluation of end of treatment treatment circulating human papillomavirus deoxyribonucleic acid (ctHPVDNA) detectability as a marker of risk of progression | Up to 5 years
  Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Functional outcomes of DART alone vs. DART + MSRT | Up to 5 years
  Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Feasibility of DART regimen outside of Mayo Clinic | Up to 5 years
  Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.

OTHER OUTCOMES:
ctHPVDNA detectability | At post-operative day 1 or 2
  Due to the limited sample size, these analyses will be hypothesis generating and descriptive in nature. Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Salivary ctHPVDNA analysis for recurrence risk and surveillance | Up to 5 years
  Salivary samples will be analyzed pre-treatment, post-op, and at the time of recurrence to determine whether salivary ctHPVDNA may further inform recurrence risk and surveillance in HPV(+) oropharyngeal squamous cell carcinoma. Due to the limited sample size, these analyses will be hypothesis generating and descriptive in nature. Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Characterization of post-operative drain fluid | Up to 5 years
  We will characterize post-operative drain fluid and compare rates of detectability to blood and saliva in order with the aim to determine whether the regional drain represents a separate regional compartment for analysis. Due to the limited sample size, these analyses will be hypothesis generating and descriptive in nature. Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Quantification of pre-treatment imaging | Up to 5 years
  We will prospectively quantify pretreatment imaging for number of involved nodes, radiographic extranodal extension as it relates to pathologic findings and risk of recurrence. Due to the limited sample size, these analyses will be hypothesis generating and descriptive in nature. Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Percentage of tumor infiltrating lymphocytes (TILs) | Up to 5 years
  We will analyze within category of low intermediate, high intermediate, and high-risk patients the percentage of TILs and association with recurrence as well as differences across treatment groups. Due to the limited sample size, these analyses will be hypothesis generating and descriptive in nature. Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Assessment of integrated vs episomal HPV | Up to 5 years
  Comparison of methods of surveillance as defined by the date of diagnosis of recurrence by ctHPVDNA testing as compared to clinical examination and imaging. Sensitivity, specificity, negative predictive value, and positive predictive value of each will be reported. Measure whether HPV is integrated vs episomal for each patient and the relationship of ctHPVDNA detectability and outcomes. These analyses will be hypothesis generating and descriptive in nature. Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.
Assess Molecular Markers Using FFPE | Up to 5 years
  We will investigate molecular markers on formalin-fixed paraffin-embedded (FFPE) from primary surgical specimens. Due to the limited sample size, these analyses will be hypothesis generating and descriptive in nature. Descriptive statistics will be summarized and the exploratory data will be correlated with clinical endpoints (PFS, time-to-progression, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, we'll use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response vs. no response), we'll use logistic regression models.

CONTACTS AND LOCATIONS:
Overall Officials: David M, Routman, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials